CLINICAL TRIAL: NCT01803399
Title: A Phase I, Randomized, Partially Blinded, Placebo- and Moxifloxacin-Controlled, 4-Period Crossover Study to Evaluate the Effect of GSK1322322 on Cardiac Conduction as Assessed by 12-lead Electrocardiogram in Healthy Volunteers (PDF112166)
Brief Title: A Study to Evaluate the Effect of GSK1322322 on Cardiac Conduction as Assessed by 12-lead Electrocardiogram in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Emerging GSK1322322 pre-clinical data ID'd potentially reactive metabolites previously not seen that changed the risk: benefit profile and led to a termination
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112166
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Infections, Bacterial
Keywords: cardiac repolarization; oral; QTc; GSK1322322; antibiotic; 12-lead ECG; placebo; IV; moxifloxacin
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK1322322 1200 mg Arm (Experimental): Each subject will receive a single dose of GSK1322322 1200 mg IV over 60 minutes on Day 1 of one of the 4 treatment periods
  Interventions: Drug: GSK1322322 1200 mg
- GSK1322322 3000 mg Arm (Experimental): Each subject will receive a single dose of GSK1322322 3000 mg IV over 60 minutes on Day 1 of one of the 4 treatment periods
  Interventions: Drug: GSK1322322 3000 mg
- Placebo Arm (Placebo Comparator): Each subject will receive a single dose of GSK1322322 Placebo IV over 60 minutes on Day 1 of one of the 4 treatment periods
  Interventions: Drug: Placebo
- Moxifloxacin 400 mg Arm (Active Comparator): Each subject will receive a single dose of moxifloxacin 400 mg administered orally on Day 1 of one of the 4 treatment periods
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: GSK1322322 1200 mg — GSK1322322 will be supplied as white to slightly colored lyophilized powder 400 mg/vial for injection. Single dose of GSK1322322 1200 mg (3 vials) will be administered IV over 60 minutes
  Arms: GSK1322322 1200 mg Arm
Drug: GSK1322322 3000 mg — GSK1322322 will be supplied as white to slightly colored lyophilized powder 400 mg/vial for injection. Single dose of GSK1322322 3000 mg (8 vials) will be administered IV over 60 minutes
  Arms: GSK1322322 3000 mg Arm
Drug: Placebo — Placebo will be supplied as 0.9% sodium chloride solution. Single dose of placebo will be administered IV over 60 minutes
  Arms: Placebo Arm
Drug: Moxifloxacin — Moxifloxacin will be supplied as oblong, dull red film coated tablets of 400 mg strength. Single dose of moxifloxacin 400 mg will be administered orally
  Arms: Moxifloxacin 400 mg Arm

SUMMARY:
This is a randomized, partially-blinded, placebo and moxifloxacin-controlled, single dose, 4-period, balanced crossover study. The primary objective of this study is to separately assess the effects of a therapeutic and supratherapeutic dose of GSK1322322 on the cardiac conduction (corrected QT interval [QTc]) compared with placebo in eligible healthy male and female subjects. Avelox (moxifloxacin hydrochloride) will be used as an open-label positive control in order to validate the sensitivity of the study in detecting QTc change. Approximately 56 healthy subjects will participate in the study for approximately 9 weeks i.e. 30 day Screening period, 4-week Treatment period, and a 7-10 day Follow-up period. There will be 4 treatment periods separated by at least 1 week. Subjects will be admitted to the clinical unit on Day -1 of each dosing period. Each subject will receive each of the four treatment sequences (GSK1322322 1200 milligram [mg] intravenous [IV] over 60 minutes x 1 dose, GSK1322322 3000 mg IV over 60 minutes x 1 dose, GSK1322322 Placebo IV over 60 minutes x 1 dose, moxifloxacin 400 mg administered orally x 1 dose) on Day 1 of each Treatment period in a randomized fashion. Twelve-lead electrocardiogram (ECG), continuous Holter monitoring, laboratory tests, vital sign measurements, and serial pharmacokinetic samples will be collected for up to 24 hours following each treatment. If no clinically significant abnormalities are noted, subjects will be discharged from the clinical research unit after the completion of all assessments on Day 2 in each period and return approximately one week later for the next dosing period. Each individual subject will follow the same dosing schedule at every period. A Follow-up visit will be conducted 7-10 days after administration of the last dose of study medication in treatment period 4.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female (of non childbearing potential) between 18 and 65 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 milli international units [mIU]/millilitre [mL] and estradiol <40 picograms [pg]/mL or <147 picomole [pmol]/litre [L] is confirmatory)
* Male subjects with female partners of child-bearing potential must agree to use one of the following contraception methods from the time of the first dose of study medication until the final follow up visit - Condom plus partner use of a highly effective contraceptive; Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Body weight >=50 kilograms (kg) for men and >=45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/(square metre) m^2 (inclusive)
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening and check-in (repeat allowed at check-in only)
* Serum Potassium, Calcium and Magnesium lab parameters within normal limits at screening and check-in (repeat allowed at check-in only)
* QTcB <450 milliseconds (msec) at screening and check-in
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* History/evidence of any arrhythmia (for example, first, second or third degree heart block, atrial fibrillation, supraventricular tachycardia, sinus bradycardia, junctional rhythm) or clinically significant cardiac disease or procedure(mitral valve regurgitation, heart murmur, angina/ischemia, congenital heart abnormalities, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA). Personal or family history of long QT syndrome
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, inflammatory bowel disease or pancreatitis. Subjects with active peptic ulcer disease or a history of upper gastrointestinal bleeding
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody result, or a positive test for Human Immunodeficiency Virus (HIV) antibody within 3 months of screening
* A positive pre-study drug/alcohol screen
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety due to potential drug interaction
* History of sensitivity to any of the study medications, quinolone antibiotics, (including moxifloxacin), or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive (serum or urine) Human chorionic gonadotropin (hCG) test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice (and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices) from 7 days prior to the first dose of study medication
* Exclusion criteria for screening Holter and ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute (bpm) for males or <50 and >100 bpm for females; PR Interval <120 and >220 msec; QRS duration <70 and >120 msec; QTc interval (Bazett) >=450 msec (Note: The waveforms must enable the QT interval to be clearly defined); Q wave >30 msec
* Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization)
* Any conduction abnormality (including but not specific to left or right bundle branch block, Atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Fridericia's formula (QTcF) for GSK1322322 as compared with time-matched placebo | Day 1: -1.5, -1.0 and -0.5 hours pre-dose (average as baseline) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose (Day 2) of each treatment period
  Triplicate 12-lead Holter ECG measurements for each subject at each time point will be averaged

SECONDARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Bazett's formula (QTcB), Individual (linear) QT correction (QTci), QT, and heart rate (HR) | Day 1: -1.5, -1.0 and -0.5 hours pre-dose (average as baseline) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose (Day 2) of each treatment period
  To estimate the effect of single dose IV GSK1322322 (1200 mg and 3000 mg) as compared with placebo. Triplicate 12-lead Holter ECG measurements for each subject at each time point will be averaged
Change from baseline in QTcB, QTci, QT, and HR | Day 1: -1.5, -1.0 and -0.5 hours pre-dose (average as baseline) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose (Day 2) of each treatment period
  To estimate the effect of single dose oral moxifloxacin (400 mg) as compared to placebo. Triplicate 12-lead Holter ECG measurements for each subject at each time point will be averaged
Plasma concentrations and selected pharmacokinetic (PK) parameters of moxifloxacin | Day 1: 15 minutes pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose (Day 2) of each treatment period
  PK parameters will include: maximum observed plasma concentration (Cmax); time to Cmax (tmax); area under the plasma concentration-time curve (AUC): from time zero (pre-dose) to last time of quantifiable concentration [AUC (0-t)], from time zero (pre-dose) to 24 hours [AUC (0-24)], and from time zero (pre-dose) extrapolated to infinite time [AUC (0-∞)]; apparent terminal phase half-life (t1/2); Systemic clearance of parent drug (CL); and volume of distribution at steady state (Vss), as data permit
Plasma concentrations and selected PK parameters of GSK1322322/moxifloxacin | Day 1: 15 minutes pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, and 24 hours post-dose (Day 2) of each treatment period
  To characterize the PK/pharmacodynamics (PD) relationship between GSK1322322/moxifloxacin plasma concentrations (and other PK parameters, if appropriate) and QTcF, QTcF changes relative to placebo (ddQTcF) , QTcB, and QTci
Safety and tolerability of GSK1322322 as assessed by change from baseline in 12-lead ECGs | Screening, Day 1 (pre-dose (x3) [mean value as baseline] and 0.5, 1, 1.5, 4, 8, 12 hours post-dose) of each treatment period, and Week 9
  Single 12-lead ECGs will be obtained
Safety and tolerability of GSK1322322 as assessed by change from baseline in vital signs | Screening, Day 1 (pre-dose (x3) [mean value as baseline] and 0.5, 1, 1.5, 4, 8, 12 hours post-dose) of each treatment period, and Week 9
  Vital sign measurements will include systolic and diastolic blood pressure, temperature and HR
Safety and tolerability of GSK1322322 as assessed by number of subjects with adverse events | Through 9 weeks
Safety and tolerability of GSK1322322 as assessed by change from baseline in toxicity grading of clinical laboratory tests | Through 9 weeks
  Clinical laboratory tests will include clinical Chemistry, hematology and urinalysis assessments

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline